CLINICAL TRIAL: NCT06436170
Title: Radial Peripapillary Vessel Density as a New Biomarker in Irvine-Gass Syndrome
Brief Title: The Role of Radial Peripapillary Vessel Density in Irvine-gass Syndrome
Acronym: OCTA and PMCE
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 05809852 Federico II
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Cataract; Macular Edema
Keywords: OCTA;RPC; IGS;PCME
MeSH Terms: conditions — Cataract; Macular Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 30 patiens with IGS mean age 70 ±6
  Interventions: Diagnostic Test: OCTA
- 30 healthy controls mean age 70 ±5
  Interventions: Diagnostic Test: OCTA

INTERVENTIONS:
Diagnostic Test: OCTA — OCTA is a non invasive diagnostic technique to visualize RPC

SUMMARY:
Pseudophakic cystoid macular edema (PCME), also known as Irvine-Gass syndrome (IGS), is an accumulation of fluid in the macula that occurs after cataract surgery, with an early or late presentation (cut-off 3 months) . It is the most common cause of decreased vision after uneventful phacoemulsification, with a rare incidence of 0.1-2.35% for clinically significant PCME .

Macular edema in IGS can be diagnosed and classified by optical coherence tomography (OCT), which enables its morphologic assessment. Fluorescein angiography (FA) is the gold standard to perform differential diagnosis for macular edema.

To date, OCT angiography (OCTA) has been proposed to study various retinal vascular diseases. In contrast to FA, OCTA is able to visualize Radial peripapillary vessel density (RCP).

The aim of this study was to investigate abnormalities in the vascular network of the optic nerve head in patients with IGS compared to healthy eyes, using OCT-A

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of PCME Cataract surgery

Exclusion Criteria:

diabetes vein occlusion uveitis vasculitis age-related macular degeneration hereditary macular dystrophy

-

Ages: 58 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of PCME following phacoemulsification, addressed to our Unit, were enrolled in the study. The diagnostic criteria for PCME were: 1) vision loss in the operated eye within 3 months after surgery in patients with acute PCME and after 3 months for patients with chronic PCME; 2) changes on B-scan structural OCT with intraretinal cystoid spaces and central macular thickness (CMT) of at least 300 micron; 3) leakage and pooling of dye in macular cystoid spaces and late hyperfluorescence of the optic nerve head on FA. Clinical suspicion of PCME was confirmed using FA and structural OCT.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
the role of OCTA in diagnosis of IGS | 10 months
  To evaluate the vascolarization of RPC in IGS

CONTACTS AND LOCATIONS:
Locations (1):
- University Federico II of Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided